CLINICAL TRIAL: NCT06686966
Title: Clinical Study on the Effect of Environmental Pollution on the Prognosis of Gastric Cancer
Brief Title: The Effect of Environmental Pollution on the Prognosis of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: ZZ2024-292-01
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancers
Keywords: gastric cancer; air pollution; environment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: gastric cancer — be diagnosed as gastric cancer

SUMMARY:
Gastric cancer is one of the common malignant tumours worldwide, with a high incidence especially in East Asia. Although the occurrence of gastric cancer is closely related to genetic factors, lifestyle and dietary habits, in recent years, environmental pollution, especially air pollution, has received more and more attention as a potential carcinogenic factor. Numerous studies have shown that harmful substances in the air such as including passive smoking, soot and oil smoke exposure, incense burning exposure, occupational exposure and outdoor work, PM2.5, PM10, nitrogen oxides, sulphur dioxide, etc. may not only induce the occurrence of gastric cancer, but also affect the prognosis of gastric cancer patients. This experiment intends to determine the extent of the influence of air pollution on the prognosis of gastric cancer by analysing the survival data of gastric cancer patients in areas with different pollution levels. In addition, the association between air pollution levels and postoperative recurrence in gastric cancer patients was investigated to find possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years;
* patients diagnosed with gastric cancer by pathological biopsy before surgery;
* patients without chemotherapy, radiotherapy, targeted and immunotherapy before enrolment;
* willing to participate in this study and sign the informed consent;
* complete clinical data.

Exclusion Criteria:

* patients with other primary malignant tumours other than gastric cancer;
* patients with systemic diseases such as severe cardiopulmonary insufficiency that affect the choice of treatment plan;
* patients who are not suitable for enrolment as assessed by the investigator;
* incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastric cancer and undergoing radical gastric cancer surgery at the First Hospital of Chongqing Medical University, the Second Hospital of Chongqing Medical University, and the Yongchuan Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
the incidence of gastric cancer | From 18 years old until the developing gastric cancer, through study completion, an average of 5 year.
  the diagnosis time of gastric cancer

IPD SHARING:
Plan to Share IPD: No
None of the three clinical centres conducting the study allowed the disclosure of patient information and data sharing.